CLINICAL TRIAL: NCT03616340
Title: Efficacy of Intra-articular NSAID Versus Corticosteroid in the Treatment of Shoulder and Knee Conditions: A Randomized, Double-Blind, Prospective Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OSF Healthcare System (Other)
Responsible Party: Principal Investigator, Miguel Ramirez, Orthopaedic Surgeon, OSF Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1209087-1
Record Dates: First submitted 2018-07-31; First posted 2018-08-06 (Actual); Last update posted 2018-08-06 (Actual); Status verified 2018-07

CONDITIONS: Knee Arthritis; Shoulder Arthritis; Shoulder Impingement; Meniscus Lesion; Rotator Cuff Tear; Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Shoulder Impingement Syndrome; Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketorolac (Experimental)
  Interventions: Drug: Shoulder injection; Drug: knee injection
- Kenalog (Experimental)
  Interventions: Drug: Shoulder injection; Drug: knee injection

INTERVENTIONS:
Drug: Shoulder injection — intra articular or subacromial shoulder injection
Drug: knee injection — intra-articular knee injection

SUMMARY:
The proposed study will compare the efficacy of Triamcinolone versus Ketorolac for intra-articular injection of the knee and shoulder

DETAILED DESCRIPTION:
This study will be a randomized prospective study comparing Triamcinolone to Ketorolac for injections in the knee and shoulder for a variety of orthopedic conditions. The investigators will monitor pain relief, length of pain relief, cost, and patient satisfaction after the injections

ELIGIBILITY:
Inclusion Criteria:

* knee and shoulder arthritis
* shoulder impingement
* rotator cuff tear

Exclusion Criteria:

* chronic pain management
* allergy to NSAIDs or steroids
* prior surgery
* kidney disease that would preclude NSAID administration

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Pain level: VAS score | 0-6 months
  VAS score
length pain relief | 0-6 months
  length of time patient reports pain relief

IPD SHARING:
Plan to Share IPD: No